CLINICAL TRIAL: NCT01458158
Title: The Role of Matrix Metalloproteinases -2 and -9 in Atherosclerosis of Patients With Chronic Kidney Disease
Brief Title: Matrix Metalloproteinases in Atherosclerosis of Chronic Kidney Disease
Acronym: MMACKD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Grigorios G. DIMAS, Doctor/PhD Candidate, Aristotle University Of Thessaloniki
Other Study IDs: A13749; 31-8-2010 (Other: AristotleU)
Record Dates: First submitted 2011-09-30; First posted 2011-10-24 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Diabetic Nephropathy
Keywords: Gelatinases; kidney disease; diabetes mellitus type 2
MeSH Terms: conditions — Diabetic Nephropathies; Kidney Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum and vessels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Diabetic nephropathy: Diabetic nephropathy in patients with type 2 diabetes
- chronic glomerulonephritis: chronic glomerulonephritis in patients without diabetes mellitus
- controls: participants without diabetic nephropathy and chronic glomerulonephritis

SUMMARY:
The purpose of this study is to determine whether matrix metalloproteinases are associated with atherosclerosis in the different stages of chronic kidney disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine the correlation of matrix metalloproteinases and atherosclerosis of chronic kidney disease. Patients with diabetes mellitus type 2,as a non-inflammatory leading cause of end stage renal failure and patients with chronic glomerulonephritis and similar course of proteinuria,as an inflammatory leading cause of end stage renal failure are enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease
* Diabetes mellitus type 2

Exclusion Criteria:

* Malignancy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from University Hospital AHEPA
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-10; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Association of matrix metalloproteinases with atherosclerosis in patients with chronic kidney disease | two years
  Matrix metalloproteinases associated with atherosclerosis in chronic kidney disease;patients with diabetes mellitus type 2 and others with chronic glomerulonephritis.Serum levels of MMPs-2 and -9 are measured by an ELISA system.Intima Media Thickness(IMT) of carotid and femoral arteries is measured with a high resolution ultrasonography.

SECONDARY OUTCOMES:
Matrix metalloproteinases and atherosclerosis associated with pro-inflammatory and oxidative stress markers in chronic kidney disease | two years
  Matrix metalloproteinases associated with atherosclerosis markers,pro-inflammatory markers and markers of oxidative stress in chronic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: Grigorios G. Dimas, MD, Principal Investigator — AHEPA University Hospital,Medical School of Aristotle University of Thessaloniki
Locations (1):
- AHEPA University Hospital, Medical School of Aristotle University of Thessaloniki, Thessaloniki, Greece